CLINICAL TRIAL: NCT00396747
Title: Phase IV Study of Early RA: a Randomized Magnetic Resonance Imaging Study Comparing the Effects of Methotrexate Alone or in Combination With Infliximab or Intravenous Pulse Methylprednisolone
Brief Title: A Comparison of Methotrexate Alone or Combined to Infliximab or to Pulse Methylprednisolone in Early Rheumatoid Arthritis: A Magnetic Resonance Imaging Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIERA
Record Dates: First submitted 2006-11-06; First posted 2006-11-07 (Estimated); Last update posted 2007-10-19 (Estimated); Status verified 2007-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Early rheumatoid arthritis,; glucocorticoids,; pulse therapy,; infliximab,; TNF blockade
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab; Methylprednisolone; Methotrexate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Active Comparator): Methotrexate
  Interventions: Drug: Infliximab, methylprednisolone, methotrexate; Drug: Methotrexate
- B (Active Comparator): MTX + MP
  Interventions: Drug: Infliximab, methylprednisolone, methotrexate; Drug: Methotrexate + Methylprednisolone
- C (Active Comparator): MTX + IFX
  Interventions: Drug: Infliximab, methylprednisolone, methotrexate; Drug: Methotrexate + Infliximab

INTERVENTIONS:
Drug: Infliximab, methylprednisolone, methotrexate
Drug: Methotrexate
  Arms: A
Drug: Methotrexate + Methylprednisolone
  Arms: B
Drug: Methotrexate + Infliximab
  Arms: C

SUMMARY:
The purpose of the study is to compare the effects of methotrexate (MTX) alone or in combination with intravenous (IV) methylprednisolone (MP) or infliximab (IFX) on MRI-detected synovitis, bone edema and erosive changes in early rheumatoid arthritis (RA) patients.

DETAILED DESCRIPTION:
The effects of Glucocorticoïds and Infliximab have never been compared in early RA using MRI as primary outcome measure. In the current study, we compare the effects of MTX alone or in combination with intravenous (IV) methylprednisolone (MP) pulse therapy or IFX on MRI-detected synovitis, bone edema and erosive changes in early RA patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible for this study if they met the American Rheumatism Association classification criteria for RA (9), had a disease duration inferior to one year, suffered from active disease (defined as the presence of a swollen joint count [SJC] ≥ 6 [by the 66 joints count] and a tender joint count [TJC] ≥ 8 [by the 68 joints count]) and had not been treated with MTX before.
* Patients were eligible for this study if they met the American Rheumatism Association classification criteria for RA (9), had a disease duration inferior to one year, suffered from active disease (defined as the presence of a swollen joint count [SJC] ≥ 6 [by the 66 joints count] and a tender joint count [TJC] ≥ 8 [by the 68 joints count]) and had not been treated with MTX before.

Exclusion Criteria:

* Exclusion criteria included past/current history of tuberculosis, congestive heart disease, past treatment with GC for more than 3 months (and not during the 4 weeks before inclusion), previous treatment with more than 2 DMARDs, MTX, IV MP pulse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2003-06; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
MRI synovitis, bone edema and erosions score | baseline, week 18 and 52

SECONDARY OUTCOMES:
Efficacy (DAS Score, ACR response) | every 2 months
Side effects | every visit

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Durez, MD, Principal Investigator — Université Catholique de Louvain
Locations (1):
- Université catholique de Louvain, Brussels, Belgium

REFERENCES:
- [Derived] Durez P, Malghem J, Nzeusseu Toukap A, Depresseux G, Lauwerys BR, Westhovens R, Luyten FP, Corluy L, Houssiau FA, Verschueren P. Treatment of early rheumatoid arthritis: a randomized magnetic resonance imaging study comparing the effects of methotrexate alone, methotrexate in combination with infliximab, and methotrexate in combination with intravenous pulse methylprednisolone. Arthritis Rheum. 2007 Dec;56(12):3919-27. doi: 10.1002/art.23055. PMID 18050189